CLINICAL TRIAL: NCT02433795
Title: A Phase II Study of Bendamustine Plus Rituximab (BR) in Patients With Relapsed or Progressive Marginal Zone B-cell Lymphoma (MZBCL)
Brief Title: Bendamustine Plus Rituximab (BR) for Relapsed or Progressive Marginal Zone B-cell Lymphoma (MZBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gyeongsang National University Hospital (Other); Korea Cancer Center Hospital (Other); Seoul National University Boramae Hospital (Other); Hallym University Medical Center (Other); Inje University (Other); Gangnam Severance Hospital (Other); Chonbuk National University Hospital (Other); Chungnam National University (Other); The Catholic University of Korea (Other); Wonju Severance Christian Hospital (Other); Gachon University Gil Medical Center (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY14-09
Record Dates: First submitted 2015-04-05; First posted 2015-05-05 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Marginal Zone B-cell Lymphoma
Keywords: Marginal zone B-cell lymphoma; bendamustine plus rituximab
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine plus rituximab(BR) (Experimental): Intravenous bendamustine plus rituximab intravenously at 1st cycle and subcutaneously from 2nd cycle (to maximum 8th cycle).
  Interventions: Drug: bendamustine plus rituximab

INTERVENTIONS:
Drug: bendamustine plus rituximab — Bendamustine 90mg/m2 IV on days 1-2 up to 6th cycle Rituximab 375mg/m2 IV on day 1 at 1st cycle Rituximab 1400mg SC on day 1 from 2nd cycle every 4 weeks up to 8th cycle

SUMMARY:
This study will be conducted to evaluate the efficacy of Bendamustine Plus Rituximab (BR) in patients with relapsed or progressive Marginal Zone B-cell Lymphoma (MZBCL).

DETAILED DESCRIPTION:
Multi-center trial, Phase II, non-randomized, open-label, single-arm study with combined therapy of bendamustine and rituximab in patients with MZBCL who has relapsed or progressive to prior chemotherapy or chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20-positive nodal or extranodal MZBCL
2. MZBCL patients who relapsed or progressed:

   * At least one and a maximum of four prior lines of chemotherapy
   * During or after the last chemotherapy or radiotherapy or
   * Without progression within 6 months of the last dose of rituximab-based regimen
3. Patients age ≥ 18 years
4. ECOG PS 0-2
5. At least one bidimensionally measurable disease
6. Adequate hematologic, renal, and hepatic functions
7. Women of child-bearing potential should use two appropriate methods of contraception during the study
8. Written informed consent

Exclusion Criteria:

1. Not all of the above inclusion criteria are met.
2. Prior chemotherapy within 4 weeks or radiotherapy within 6 weeks
3. Corticosteroids during last 28 days except chronic administration of prednisolone at a dose of < 20mg/day for indications other than lymphomas
4. Evidence of CNS involvement by lymphomas
5. Active HBV/HCV infections, known HIV infection
6. Prior diagnosis of cancers within 5 years, except cervical intraepithelial neoplasia type 1, localized non-melanoma skin cancer, or small differentiated thyroid cancer
7. Serious concurrent disease:
8. Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate based on Revised Response Criteria for Malignant Lymphoma | 6 months

SECONDARY OUTCOMES:
Complete remission rate | 6 months
Safety based on NCI CTCAE version 4.0 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dae Seog Heo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (11):
- South Korea (11):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Hallym University Medical Center, Anyang-si
  - Chungnam National University, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - Inje Universit, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul